CLINICAL TRIAL: NCT03347617
Title: Response Assessment to Pembrolizumab With Standard of Care Therapy in Glioblastoma Using Ferumoxytol Steady State Imaging- A Pilot Study
Brief Title: Ferumoxytol MRI in Assessing Response to Pembrolizumab in Patients With Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator transition
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Leslie Muldoon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016046; NCI-2017-02008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016046 (Other: OHSU Knight Cancer Institute); K08CA237809 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-20 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Ferumoxytol MRI, pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 years or 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive ferumoxytol IV and undergo MRI scans at baseline, 4 weeks after the last day of standard of care stereotactic radiosurgery or chemoradiotherapy, every 9 weeks thereafter until suspected radiographic progression, and then within 4 weeks from suspected radiographic progression.
  Interventions: Drug: Ferumoxytol; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo ferumoxytol MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This pilot phase II trial studies how well ferumoxytol magnetic resonance imaging (MRI) works in assessing response to pembrolizumab in patients with glioblastoma. Diagnostic procedures, such as ferumoxytol MRI, may help measure a patient's response to pembrolizumab treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the sensitivity and specificity of relative cerebral blood volume (rCBV) measured by steady state MRI with ferumoxytol in identifying true versus (vs) pseudoprogression in patients with newly diagnosed glioblastoma multiforme (GBM) receiving pembrolizumab with standard of care chemo-radiation.

SECONDARY OBJECTIVES:

I. Determine the safety and toxicity of pembrolizumab when used in combination with standard of care chemo radiation.

II. Determine the progression free survival (PFS), overall survival (OS), clinical response and duration of best response.

EXPLORATORY OBJECTIVES:

I. Compare the immune response as determined by the volume, pattern and intensity of delayed (24 hour [hr]) ferumoxytol uptake between subjects who develop true vs pseudoprogression.

II. Investigate the serum immunological parameters (serum biomarker) and correlate clinical as well as radiological response with systemic immune response to pembrolizumab as measured by immunological panel.

III. Compare the changes in PDL-1 expression in the biopsy tissue before and after therapy at the time of progression and correlate PD-L1 expression with response rates and survival.

IV. Investigate the feasibility of measuring vascular volume fraction (VVF), vessel size index (VSI) and vessel density index (VDI) as surrogate for response (true vs pseudoprogression, as determined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 and immune related response criteria [irRC]).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 years or 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive ferumoxytol IV and undergo MRI scans at baseline, 4 weeks after the last day of standard of care stereotactic radiosurgery or chemoradiotherapy, every 9 weeks thereafter until suspected radiographic progression, and then within 4 weeks from suspected radiographic progression.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for up to 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have a life expectancy of at least 6 months
* Have a histologically confirmed diagnosis of:

  * Newly diagnosed glioblastoma (World Health Organization [WHO] grade IV)
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 on stable or reducing dose of steroids for symptom management (not more than 8 mg of dexamethasone or equivalent per day) for 5 days prior to enrollment; change in glucocorticoid dose for any purpose other than to modulate symptoms from an adverse event; Note: The use of physiologic doses (e.g., prednisone 10 mg) of corticosteroids may be approved after consultation with Merck & Co; use of prophylactic corticosteroids to avoid allergic reactions (e.g. IV contrast dye) is permitted
* At least 14 days from any major surgeries including brain biopsy before the start of study drug pembrolizumab
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; male subjects should agree to use an adequate method of contraception, including but not limited to, abstinence from heterosexual activity starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Subject is eligible for and agrees to receive standard of care radiation and temozolamide after biopsy or maximum safe surgical resection

Exclusion Criteria:

* Has a diagnosis of immunodeficiency including human immunodeficiency virus (HIV) (HIV 1/2 antibodies) and is not on continuous daily immunosuppressive therapy within 7 days prior to the first dose of trial treatment; (an exception to this is the use of steroids for brain edema and resulting symptom); subjects may receive a stable or reducing dose of steroids (up to 8 mg dexamethasone or equivalent for at least 5 days prior to signing consent) to prevent or manage cerebral edema; subjects requiring over 8mg of dexamethasone per day on or five days prior to signing consent are excluded)
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or ferumoxytol or any of their excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2009); subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who have a contraindication for 3T MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated
* Subjects with known iron overload (genetic hemochromatosis); in subjects with a family history of hemochromatosis, hemochromatosis must be ruled out prior to study entry with normal values of the following blood tests: transferrin saturation (TS) test and serum ferritin (SF) test; all associated costs will be paid by the study
* Subject who have received ferumoxytol within 3 weeks of study entry
* Subjects with three or more drug allergies from separate drug classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Muldoon, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Started | 52
Completed (Completed is defined as completing at least one evaluable study imaging session after radiation.) | 43
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 51
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Specificity of Identifying Pseudoprogression
Description: Sensitivity and specificity are measures for the diagnostic performance of rCBV (relative cerebral blood volume) to distinguish between pseudoprogression and true progression. Sensitivity measures how well Fe-SS-rCBV identifies those who have true progression, and specificity those who have psuedoprogression. Because rCBV is a continuous variable, the cutoff point for this analysis was 1.75.
Time Frame: At suspected progression, up to two years.
Population: A total of 12 out of 52 participants were evaluable to allow calculation of specificity to distinguish true progression from pseudo-progression based on steady state rCBV at suspected progression
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Diagnostic (Ferumoxytol MRI, Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 years or 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive ferumoxytol IV and undergo MRI scans at baseline, 4 weeks after the last day of standard of care stereotactic radiosurgery or chemoradiotherapy, every 9 weeks thereafter until suspected radiographic progression, and then within 4 weeks from suspected radiographic progression.
  Ferumoxytol: Given IV Laboratory Biomarker Analysis: Correlative studies Magnetic Resonance Imaging: Undergo ferumoxytol MRI Pembrolizumab: Given IV
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 12
percentage | 58.3 [27.9 to 84.8]

2. Primary Outcome: Sensitivity of Identifying True Progression
Description: The calculation of sensitivity is based on steady state rCBV (relative cerebral blood volume) at suspected progression. Cutoff point 1.75.
  Sensitivity and specificity are measures for the diagnostic performance of rCBV (relative cerebral blood volume) to distinguish between pseudoprogression and true progression. Sensitivity measures how well Fe-SS-rCBV identifies those who have true progression, and specificity those who have psuedoprogression. Because rCBV is a continuous variable, the cutoff point for this analysis was 1.75.
Time Frame: At suspected progression, up to two years.
Population: A total of 15 out of 52 participants were evaluable to allow calculation of sensitivity to distinguish true progression from pseudo-progression based on steady state rCBV at suspected progression
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 15
percentage | 46.7 [21.3 to 73.4]

3. Secondary Outcome: Progression Free Survival
Description: Will be assessed using the Kaplan-Meier product limit estimates. Response assessment was completed based on a modified version of the Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: Until off study, up to 5 years.
Population: All enrolled subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 52
Months | 10.4 [7.1 to 11.7]

4. Secondary Outcome: Overall Survival
Description: Will be assessed using the Kaplan-Meier product limit estimates.
Time Frame: Until off study, up to 5 years.
Population: All enrolled subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 52
Months | 15.2 [12.5 to 17.1]

5. Secondary Outcome: Duration of Best Response
Description: Will be analyzed using the Kaplan-Meier product limit estimates. Response assessment was completed based on a modified version of the Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: Until off study, up to 5 years.
Population: All enrolled subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 52
Months | 6.4 [4.1 to 8.5]

6. Secondary Outcome: Disease Response
Description: Disease response was assessed based on a modified version of the Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: Until off study, up to 5 years.
Population: Of the 52 enrolled patients, 43 were evaluable (9 replaced).
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 43
Participants
  Complete response | 8
  Partial response | 18
  Stable disease | 9
  Disease progression | 8

7. Secondary Outcome: Determine the Safety and Toxicity of Pembrolizumab When Used in Combination With Standard of Care Chemo Radiation.
Description: Number of participants with adverse events possibly related or related to pembrolizumab in combination with standard of care. Will be analyzed using proportions and exact 95% confidence intervals.
Time Frame: 30 days after last dose of pembrolizumab, up to 2 years.
Population: Out of 52 participants, 29 experienced an adverse event greater than or equal to grade 3 that were possibly related or related to pembrolizumab.
Measure: Number; unit: participants
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
Number analyzed (Participants) | 52
participants
  Grade 3 or above possibly related to pembrolizumab | 27
  Grade 3 or above related to pembrolizumab | 2

ADVERSE EVENTS:
Time Frame: All AEs were recorded up to 30 days after last pembrolizumab (maximum treatment of pembrolizumab is 2 years) except all-cause mortality which was monitored/assessed for up to 5 years.
Arm/Group | Diagnostic (Ferumoxytol MRI, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 45/52
Serious Adverse Events (participants affected / at risk) | 15/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic (Ferumoxytol MRI, Pembrolizumab) (N=52)
Myocardial infarction (Cardiac disorders) | 1
Flu like symptoms (General disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 3
Thromboembolic event (Vascular disorders) | 1
Edema cerebral (Nervous system disorders) | 2
Nausea/vomiting (Gastrointestinal disorders) | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 1
Seizures (Nervous system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Pleocytosis (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hypotension (Vascular disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 1
Wound infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 1
Psychiatric disorders - Other, specify - altered mental status (Psychiatric disorders) | 1
Eye lid function disorder - drooping (Eye disorders) | 1
Gait disturbance (General disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic (Ferumoxytol MRI, Pembrolizumab) (N=52)
Anemia (Blood and lymphatic system disorders) | 24
CD4 lymphocytes decreased (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 9
Lymphocyte count decreased (Blood and lymphatic system disorders) | 41
Neutrophil count decreased (Blood and lymphatic system disorders) | 5
Platelet count decreased (Blood and lymphatic system disorders) | 31
White blood cell decreased (Blood and lymphatic system disorders) | 6
Ear pain (Ear and labyrinth disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 4
Hyperthyroidism (Endocrine disorders) | 5
Hypothyroidism (Endocrine disorders) | 6
Blurred vision (Eye disorders) | 11
Other eye disorders (Eye disorders) | 5
Alanine aminotransferase increased (Gastrointestinal disorders) | 25
Alkaline phosphatase increased (Gastrointestinal disorders) | 9
Anorexia (Gastrointestinal disorders) | 10
Aspartate aminotransferase increased (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 30
Stomach pain (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 7
Edema (General disorders) | 6
Fatigue (General disorders) | 38
Fever (General disorders) | 5
Localized edema (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Weight loss (General disorders) | 3
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 8
Bruising (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 20
Hypernatremia (Metabolism and nutrition disorders) | 4
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 14
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 5
LDH increased (Metabolism and nutrition disorders) | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Ataxia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 11
Dysarthria (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Gait disturbance (Nervous system disorders) | 9
Headache (Nervous system disorders) | 26
Memory impairment (Nervous system disorders) | 19
Nervous system disorders - Other, specify (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 12
Tremor (Nervous system disorders) | 4
Agitation (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 11
Confusion (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Hematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 6
Thromboembolic event (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03347617/Prot_SAP_000.pdf